CLINICAL TRIAL: NCT04623970
Title: Çocuk Hastalarda Değişik Konsantrasyonlarda Kullanılan Sedasyon Ajanlarının Anksiyete Üzerine Etkilerinin Değerlendirilmesi
Brief Title: Evaluation of the Effects Using the Combination of Sedative Agents on Dental Anxiety in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, volkan Ciftci, Director, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 82/2
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Anxiety Postoperative
Keywords: Dental anxiety; Deep Sedation; Ketofol; Propofol; Salivary Cortisol
MeSH Terms: interventions — Dental Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol sedation group (Experimental): Patients in this experimental group received propofol sedation agent.
  Interventions: Procedure: Dental Treatment
- Ketofol 1:3 sedation group (Experimental): Patients in this experimental group received ketofol sedation agent as a 1:3 mixture.
  Interventions: Procedure: Dental Treatment
- Ketofol 1:4 sedation group (Experimental): Patients in this experimental group received ketofol sedation agent as a 1:4 mixture.
  Interventions: Procedure: Dental Treatment

INTERVENTIONS:
Procedure: Dental Treatment — Comprehensive dental care (restorative treatmen, crowns, pulp therapy, fissure sealant and teeth extraction for pediatric patients under the deep sedation

SUMMARY:
The aims of this study were firstly, to evaluate the changes in the anxiety level after deep sedation with various intravenous sedative agents using salivary cortisol level in pediatric dental patients and secondly, to compare clinical effectiveness of this sedative agents, perioperative complications, recovery time and adverse effects.

DETAILED DESCRIPTION:
This clinical study was included 69 healthy pediatric patients aged 3 to 7 years with high anxiety. The patients were divided into 3 groups according to the sedative agents: Group 1 (n=23) was received Propofol, Group 2 (n=23) was receieved Ketofol 1:3, and Group 3 (n=23) was received Ketofol 1:4. The anxiety levels were assessed using Facial Image Scale (FIS) anxiety scale and changes in salivary cortisol levels were assessed using ELISA before and after the drug administration. Perioperative vital signs, depth of sedation were recorded at intervals of 5 minutes. Preoperative and postoperative complications, operation and recovery time were recorded in the follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients age between 3-7 years old
* Having no systemic condition and ASA 1 healty status
* Having high dental anxiety
* Having no dental treatment under the sedation or general anesthesia before
* Having no dental treatment before

Exclusion Criteria:

* Having obstructed nasal passages, raised intracranial or intraocular pressure, allergy
* Using any drug which effected saliva construction
* Having enough saliva for saliva cortisol evaluation

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — 35 Male and 34 Female
Enrollment: 69 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Dental anxiety (subjective) | through study completion, an average of 12 months
  Units on a Scale (Patient's dental anxiety level was evaluated with Facial Image Scale after treatment. Patients signed from 1 to 5 score for dental anxiety.The data were collected and statistically analysed using by the numerical data. In this study, "1" and "2" scores are considered as better outcome. Patients who signed these scores described as no anxiety. The worst outcome is considered as the patients signed "4-5". Each scale range for each time interval evaluated as count of patient and presented as percentage.)
Dental anxiety (objective) | through study completion, an average of 12 months
  Units on Saliva cortisol levels (Dental anxiety was evaluated with Enzyme-linked immunosorbent assay after treatment.The patients were measured from 0 to 200 nmol/L for dental anxiety after the treatment.The data were collected and statistically analysed using by the numerical data. In this study, " 0-28 nmol/L'' are considered as better outcome. Patients who were have these scores described no dental anxiety for deep sedation. The worst outcome is considered as the anxious patients have ">28 nmol/L ". Each value range for each time interval evaluated as count of patient and presented as percentage.)
Depth of sedation | through study completion, an average of 12 months
  Units on a Scale (Depth of sedation was evaluated with Ramsay Sedation Scale during the sedation. Observer signed from 0 to 5 score for depth of sedation during the treatment.The data were collected and statistically analysed using by the numerical data. In this study, "4-5" scores are considered as better outcome. Patients who were signed these scores described as sedated patients for dental treatment. The worst outcome is considered as the patients signed "0-3". Each scale range for each time interval evaluated as count of patient and presented as percentage.)
Postperative complications | through study completion, an average of 12 months
  Units on a Scale ( Postoperative complications were evaluated with a form which was included absence or presence of agitation, hypersalivation, nausea-vomiting and double vision. Observer signed absence or presence for each complications after the treatment.The data were collected and statistically analysed using by the numerical data)
Perioperative complications | through study completion, an average of 12 months
  Units on a Scale (Perioperative complications were evaluated with a form which was included absence or presence of local injection pain, cough, saturation drop and spontaneous movement. Observer signed absence or presence for each perioperative complications during the deep sedation.The data were collected and statistically analysed using by the numerical data)

SECONDARY OUTCOMES:
Heart Rate | through study completion, an average of 12 months
  Differents Units of measure (Heart rate beats in bpm was measured per five minutes during the operation)
Systolic and diastolic arterial pressure | through study completion, an average of 12 months
  Differents Units of measure (Systolic and diastolic arterial pressures in mmHg were measured per five minutes during the operation)
Oxygen saturation | through study completion, an average of 12 months
  Differents Units of measure (Oxygen saturation in mmHg was measured per five minutes during the operation)

CONTACTS AND LOCATIONS:
Overall Officials: volkan Ciftci, Study Director — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)